CLINICAL TRIAL: NCT01873677
Title: A Randomized, Vehicle Controlled, Double Blind, Parallel Group, Multi Center Phase III Study to Evaluate the Safety and Efficacy of M518101 in Subjects With Plaque Psoriasis
Brief Title: Study to Evaluate the Efficacy and Safety of M518101 in Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho North America Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M518101-US02
Record Dates: First submitted 2013-06-06; First posted 2013-06-10 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (Placebo Comparator): Proper quantity twice a day
  Interventions: Drug: Vehicle
- M518101 (Experimental): Proper quantity twice a day
  Interventions: Drug: M518101

INTERVENTIONS:
Drug: M518101
  Arms: M518101
Drug: Vehicle
  Arms: Vehicle

SUMMARY:
This study is to evaluate the efficacy and safety of M518101 in subjects with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Who are able and willing to give signed informed consent
* Who are male or females aged 18 years or older with plaque psoriasis confirmed by the Investigator.
* Who have up to 20% of body surface area (BSA) afflicted with plaques
* Who are neither pregnant nor breast-feeding, nor plan to become pregnant during the study.

Exclusion Criteria:

* Who have a history of allergy to vitamin D3 derivative preparations or a history of relevant drug hypersensitivity.
* Who are pregnant or lactating.
* Who have any renal or hepatic insufficiency, or clinically significant cardiac, renal or hepatic disease.
* Who are not deemed eligible as determined by medical history, physical examination or clinical laboratory safety tests.
* Who have clinically relevant history or presence of any disease or surgical history other than psoriasis which is likely to affect the conduct of the study.
* Whose serum calcium levels exceed the upper limit of reference range
* Who have used any investigational medicinal product and/or participated in any clinical study within 60 days of randomization.
* Who have been treated with systemic therapy within 30days of randomization.
* Who have treated with biologics within 5 half-lives of the biologics before the day of randomization
* Who have been treated with topical therapy within 14days before the day of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment | 8 weeks after dosing

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Coastal Clinical Research, Mobile, Alabama
  - Omni Dermatology, Phoenix, Arizona
  - Skin Surgery Medical Group, San Diego, California
  - University Clinical Trials, San Diego, California
  - The Savin Center, New Haven, Connecticut
  - Visions Clinical Research, Boynton Beach, Florida
  - North Florida Dermatology Associates, Jacksonville, Florida
  - International Dermatology Research Inc, Miami, Florida
  - FXM Research Miramar, Miramar, Florida
  - Renstar Medical Research, Ocala, Florida
  - Belleair Research Center, Pinellas Park, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Shondra Smith Dermatology & Advanced Aesthetics, Lake Charles, Louisiana
  - Radiant Research, Edina, Minnesota
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - PMG research of Raleigh, Cary, North Carolina
  - Atlantic Dermatology Associates, Wilmington, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma University Health Science Center, Oklahoma City, Oklahoma
  - Philadelphia Institute of Dermatology, Fort Washington, Pennsylvania
  - Derm Dox Center for Dermatology, Hazleton, Pennsylvania
  - Clinical Partners, Johnston, Rhode Island
  - Rhode Island Hospital Dermatology, Providence, Rhode Island
  - Radiant Research, Greer, South Carolina
  - The Center for Skin Research, Houston, Texas
  - Suzanne Bruce and Associates The Center for Skin Research, Katy, Texas
  - Dermatology Clinical Res., San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Dermatology Associates, Seattle, Washington